CLINICAL TRIAL: NCT01914562
Title: An Open Label Trial to Assess the Effects of Food on the Pharmacokinetic Parameters of Obeticholic Acid (OCA)
Brief Title: Effect of Food on Pharmacokinetics of Obeticholic Acid (OCA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 747-104
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — obeticholic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- OCA 10 mg while fasted (Experimental): OCA 10 mg orally in the fasting state
  Interventions: Drug: OCA 10 mg
- OCA 10 mg while Fed (Experimental): OCA 10 mg orally in the fed state
  Interventions: Drug: OCA 10 mg
- OCA 25 mg while fasted (Experimental): OCA 25 mg orally in the fasting state
  Interventions: Drug: OCA 25 mg
- OCA 25 mg while Fed (Experimental): OCA 25 mg orally in the fed state
  Interventions: Drug: OCA 25 mg

INTERVENTIONS:
Drug: OCA 10 mg — OCA 10 mg tablet oral
  Other Names: 6α-ethyl chenodeoxycholic acid;(6-ECDCA), INT-747
  Arms: OCA 10 mg while Fed; OCA 10 mg while fasted
Drug: OCA 25 mg — OCA 25 mg tablet oral
  Other Names: 6α-ethyl chenodeoxycholic acid;(6-ECDCA), INT-747
  Arms: OCA 25 mg while Fed; OCA 25 mg while fasted

SUMMARY:
This is an open label, randomized, balanced, single center, single dose, trial to assess the pharmacokinetic (PK) profile of OCA, glyco-OCA and tauro-OCA on an empty stomach (fasted condition) and following a high fat, high calorie meal (fed condition) in a 2-period, 2-sequence, crossover manner.

ELIGIBILITY:
Inclusion Criteria:

Subjects are required to meet the following criteria in order to be included in the trial.

1. Male or female subjects from 18 to 55 years
2. Contraception: Female subjects must be postmenopausal, surgically sterile, or if premenopausal, be prepared to use more than 1 effective (≤ 1% failure rate) method of contraception during the trial and until at least 30 days after the last dose of OCA. Effective methods of contraception are considered to be:

   1. Double barrier method, ie, (a) condom (male or female) with spermicide or (b) diaphragm with spermicide
   2. Intrauterine device (IUD)
   3. Vasectomy
3. Good general health as determined by medical history, and by results of physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory tests obtained within 14 days prior to Day 0
4. Body mass index (BMI) of 18 to 28; BMI is determined by the following equation: BMI = weight/height2 (kg/m2).
5. Willing to abstain from alcohol, caffeine, and xanthine-containing food and beverages for 72 hours prior to each period check in and during participation of the inpatient periods of the trial
6. Willing and able to give written informed consent

Exclusion Criteria:

Subjects meeting the following criteria will be excluded from the trial.

1. Prior participation in a clinical trial of OCA (INT-747; 6-ECDCA)
2. History or presence of any disease or condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs including bile salt metabolism in the large intestine, eg, inflammatory bowel disease
3. History of gastrointestinal surgeries or gall bladder removal (cholecystectomy)
4. History or presence of a clinically significant cardiovascular, hepatic, diabetic, gastrointestinal, metabolic, neurologic, pulmonary, endocrine, psychiatric, or neoplastic disorder(s)
5. History of known or suspected clinically significant hypersensitivity to any drug, aside from penicillin
6. Ingestion of a prescription medication within 14 days prior to Day 0 or ingestion of an over the counter medication within 7 days prior to Day 0
7. Participation in radiologic examinations involving parenteral administration of iodinated contrast materials within 2 weeks prior to screening, or subsequently, through the end of trial participation
8. History or presence of alcohol abuse (defined as consumption of more than 210 mL of alcohol per week; or the equivalent of fourteen 4 ounces (oz) glasses of wine, or fourteen 12 oz cans/bottles of beer or wine coolers per week)
9. History or presence of substance abuse within the past 2 years or positive drug screen tests
10. Smoker or user of tobacco or nicotine products
11. Any screening laboratory test for which the results are not within the normal reference range and considered clinically significant
12. Participation in another investigational drug trial within 30 days prior to Day 0
13. History of noncompliance to medical regimens, or subjects who are considered to be potentially unreliable
14. Blood or plasma donation within 30 days prior to Day 0
15. Mental instability or incompetence
16. Presence of human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV) at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) - fed and fasted | Day 1 and Day 14: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, and 14 hours
  maximum concentration (observed)
Time to maximum concentration (Tmax) | 24 hours
  Time to maximum concentration
Area under the concentration versus time (AUCt) | 216 hours
  Area under the concentration versus time curve from time 0 to the last sampling time with measurable analyte concentration.
Area under the concentration versus time curve from 0 to 24 hours (AUC 0-24) | 24 hours
  Area under the concentration versus time curve from 0 to 24 hours with measurable analyte concentration

CONTACTS AND LOCATIONS:
Overall Officials: David Shapiro, MD, Study Director — Intercept Pharmaceticals, Inc.; Terry E. O'Reilly, MD, Principal Investigator — Celrion, Inc.
Locations (1):
- Celerion, Inc., Tempe, Arizona, United States